CLINICAL TRIAL: NCT02495012
Title: A Multi-centered, Randomized, Double-blinded, Placebo-Parallel Controlled Phase IIb Clinical Study to Evaluate the Safety and Efficacy of Antiplatelet Thrombolysin Injection for the Treatment of Patients With ST Segment Elevation Myocardial Infarction (STEMI) Before Receiving PCI Therapy.
Brief Title: Anfibatide Treatment in STEMI Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LeesPahrm_Anfibatide_Phase2b
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: efficacy; safety; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — agkisacucetin protein, Agkistrodon acutus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): 5IU/60 kg bolus and 0.002 IU/kg/h continuous infusion for 48 hours
  Interventions: Drug: placebo
- treatment (Active Comparator): 5IU/60 kg bolus and 0.002 IU/kg/h continuous infusion for 48 hours
  Interventions: Drug: Anfibatide

INTERVENTIONS:
Drug: placebo — Freeze-dried powder without snake venom will be dissovled in saline
  Arms: control
Drug: Anfibatide — Freeze-dried powder with snake venom will be dissovled in saline
  Arms: treatment

SUMMARY:
A Phase IIb clinical trial to investigate the safety and efficacy of antiplatelet thrombolysin injection for patients with ST Segment Elevation Myocardial Infarction (STEMI) before receiving PCI therapy, in order to provide evidence for Phase III design.

DETAILED DESCRIPTION:
Anfibatide is a snake venom, and we have investigated it in humans for many years with phase 1&2a studies. A Phase IIb clinical trial to investigate the safety and efficacy of antiplatelet thrombolysin injection for patients with ST Segment Elevation Myocardial Infarction (STEMI) before receiving PCI therapy, in order to provide evidence for Phase III design.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. Fulfill the standard of direct PCI: ST Segment Elevation Myocardial Infarction occurred < 12 hours (ST Segment Elevation or New Left Bundle Branch Block (LBBB), combined myocardial ischemia chest pain medical history or the dynamic change of cardiac marker (troponin and/or CK-MB);
3. Patients who will receive PCI and suitable for angioplasty and stent placement;
4. Patients, or their family or guardian give signed informed consent forms.

Exclusion Criteria:

1. Patients with weight < 50kg;
2. Patients with severe hepatic or renal dysfunction, alanine aminotransferase (ALT) exceeds 3 times the normal maximum reference level, creatinine clearance level < 30ml/min or serum creatinine ≥ 200μmol/L or ≥2.5mg/dl;
3. Patients with severe hemodynamic instability;
4. Patients who will receive 2 times or more PCI treatment;
5. Patients with heart function in decompensatory phase (Killip grade 3-4) or cardiac shock;
6. Patients with untreated hypertension (SBP > 180mmHg or DBP > 110mmHg) or hypotension shock (SBP < 90mmHg);
7. Patients received GPIIb/IIIa receptor antagonists and/or thrombolytic therapy before randomization;

   1. Used eptifibatide and tirofiban in the past 12 hours before the randomization;
   2. Used abxicimab in the past 7 days before the randomization;
   3. Have received thrombolytic therapy before the randomization;
8. Patients who need a long-term treatment of clopidogrel;
9. Patients who have received enoxaparin sodium injection before the surgery;
10. Patients who have hemorrhage risk:

    1. Suffered from ischemic stroke or transient ischemic attack (TIA) in the past 12 months;
    2. Suffered from hemorrhage stroke, or other life-long neuronal dysfunction;
    3. Suffered from tumor, arteriovenous malformation in brain and aneurysms;
    4. Suffered from traumatic brain injury in the past 3 months, or received major surgery;
    5. Received percutaneous coronary intervention (PCI) in the past 6 months;
    6. Have received coronary artery bypass graft therapy (CABG);
    7. Receiving long-term oral anticoagulants therapy;
    8. Suffered from active peptic ulcer, urinary and reproductive tract hemorrhage, or other active hemorrhage.
11. Patients with coagulation disorder:

    1. Known as international normalized ratio > 2*;
    2. Patients with coagulation abnormalities or other hemorrhagic tendency (including inherited hemorrhagic diseases, e.g. Von Willebrand disease or hemophilia; acquired hemorrhagic diseases; and other clinically identified hemorrhagic diseases with unsolved rationale);
    3. Hematology test shows platelet count < 100x109mm3/L, or hemoglobin < 100g/L;
    4. Recorded clopidogrel-related thrombocytopenia or agranulocytosis;
12. Life expectancy < 1 year;
13. Patients who have implemented with pacemaker, and contraindicated to MRI examination;
14. Patients who are allergic constitution or allergic to any component of aspirin, clopidogrel, creatinine, antiplatelet thrombolysin and investigational product;
15. Women in pregnant or lactation period, or women of child-bearing age do not take efficient contraception measures;
16. Patients who are participating or will be participating in other clinical trials;
17. Patients who have participated in clinical trials of antiplatelet thrombolysin or other related trials;
18. Patients who are not suitable for participating in this clinical trial according to the investigator's judgment, including who are unable or unwilling to follow the protocol;
19. Patients who participated in other clinical trials in the past 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-03 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
ratio of TMPG grade 2 and grade 3 | within 24 hours
  After PCI, TMPG grade will be evaluated and

SECONDARY OUTCOMES:
inhibition rate of platelet aggregation and GP1b receptor combination rate | 48 hours
  Baseline, 15-20 minutes after injection, 24-26 hours after injection, 48-50 hours after injection, 8-10 hours after the cease of medication, the comment and analysis of the inhibition rate of platelet aggregation and GP1b receptor combination rate
Patients ratio of no-reflow to slow-flow in coronary artery after PCI therapy | 24 hours
Analysis of iconography reference: instant TIMI, CTFC and TMPG before/after the target vessel revascularization PCI therapy | 24 hours
The depression level of ST segment from right after the PCI therapy to 2 hours later | within 24 hours
  i. Complete: depression level ≥ 70% ii. Partially: 30% ≤ depression level < 70% iii. None: < 30%
Compare the baseline troponin level to the troponin level at 24-26 hours after injection and at 3 days after the surgery respectively | 72 hours
(6) Check the CMR at 3-5 days after the surgery, evaluate the Myocardium Salvage Index (MSI) | 5 days
(7) While surgery and hospitalization, follow the ratio and dose as suggested by the surgeon in case of emergency use of GP IIb/IIIa receptor antagonist or other antiplatelet drug | 5 days
(8) Clinical endpoint 30 days after surgery (caused by death, non-fatal myocardial infarction reissue, blood clot formation after stent implantation, non-fatal stroke, target lesion revascularization reissue) and the analysis of the causes | 30days
Recorded hemorrhage issues for 30 days after the surgery (BARC hemorrhage standard) | 30days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First hospiatl, Beijing, China